CLINICAL TRIAL: NCT06760325
Title: The Effect of a Tidal Model-Based Approach Applied During Home Visits on Mental Health Parameters and Hospital Admission Frequency in COPD Patients: a Randomized Controlled Trial
Brief Title: The Effect of a Tidal Model-Based Approach Applied During Home Visits on Mental Health Parameters and Hospital Admission Frequency in COPD Patients
Acronym: Tidal Model
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kilis 7 Aralik University (Other)
Collaborators: Mersin University (Other)
Responsible Party: Principal Investigator, Özcan ÖZDEMİR, Res. Asst., Kilis 7 Aralik University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2024-OEM.1231; 2024-E.58302 (Registry Identifier: Ethics Committee Approval Number)
Record Dates: First submitted 2024-12-30; First posted 2025-01-06 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: COPD III/IV
Keywords: Tidal Model; COPD; Mental Health; Home Visits
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Interventional
Who Masked: Participant
Masking Description: Specify as needed (Single Blind)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Arm (No Intervention) (No Intervention): In this arm, Tidal Model-based approaches will not be applied during home visits to COPD patients. No psychosocial interventions were provided to patients, and standard care was maintained.
- Experimental Arm (Tidal Model Intervention) (Experimental): In this arm, Tidal Model-based psychosocial interventions will be applied during home visits to COPD patients.
  Interventions: Behavioral: Tidal Model Intervention

INTERVENTIONS:
Behavioral: Tidal Model Intervention — The model emphasizes long-term developmental care, extending support from hospital to home after discharge. This approach equips individuals with skills to understand and address challenges, emphasizing therapeutic interventions and sustained support through professionals or community groups. By focusing on the "chaos" and "tide" concepts of the Tidal Model, psychosocial interventions aim to enhance independence, manage symptoms, and improve quality of life.
  In this arm, Tidal Model-based approaches will be applied during home visits to COPD patients. Within the scope of the intervention, psychosocial needs of patients will be assessed, individualized care plans will be created and symptom management and independence will be promoted by focusing on the "chaos" and "tide" concepts of the Tidal Model.
  Arms: Experimental Arm (Tidal Model Intervention)

SUMMARY:
Despite the recent increased interest in identifying the needs of COPD patients and improving disease management, monitoring the psychosocial well-being of these individuals remains insufficient. Nursing care that incorporates psychosocial approaches plays a critical role in halting disease progression and controlling symptoms in COPD management. The Tidal Model emerges as a vital tool in enhancing patient independence throughout this process. This recovery-oriented model provides a robust framework for individualized care by thoroughly analyzing patients' needs. It likens life to an ocean voyage and emphasizes learning how to cope with challenges encountered during this journey. The difficulties experienced by individuals with chronic illness and respiratory limitations are aligned with the Tidal Model's concepts of chaos and tides.

Current studies indicate that psychological interventions for COPD patients have limited effectiveness in reducing psychological morbidity. Additionally, while interventions such as mindfulness-based and digital approaches show promise, their effects have not consistently proven significant across studies. This underscores the ongoing challenge of effectively addressing the psychological aspects of COPD and highlights the need for further research to identify more robust interventions.

In this context, guided by the philosophy of the Tidal Model that emphasizes "helping individuals with problems in living," it has been hypothesized that the model would be suitable for use with individuals with COPD. The current study aims to evaluate its effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Clinical diagnosis of COPD for at least one year
* No cognitive or sensory disabilities
* No prior participation in any psychosocial support training
* GOLD stage 'E' COPD
* Availability of a private or suitable room for interviews
* Residence within the city center

Exclusion Criteria:

* Age under 18 years
* Declined participation in the study
* Cognitive or sensory disabilities
* Prior participation in any psychosocial support training
* GOLD stage 'A' or 'B' COPD
* Unsuitable environment for conducting interviews
* Security concerns for the researcher
* Residence outside the city center or in rural areas

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2025-08-29 (Estimated)

PRIMARY OUTCOMES:
Mental Well-being Score | Assessments will be conducted at three time points: baseline, post-intervention (after 7 weeks), and at the 19-week follow-up.
  The Warwick-Edinburgh Mental Well-being Scale was developed by Tennant and colleagues (2007) to measure the mental well-being levels of individuals in the United Kingdom. Encompassing both 'psychological well-being' and 'subjective well-being', the scale consists of 14 positive items. Higher scores on the scale indicate higher levels of mental well-being. The Warwick-Edinburgh Mental Well-being Scale Short Form (WEMWBS-SF) is a 7-item scale using a 5-point Likert scale (1=Never, 5=Always) and is composed of positive statements. This study opted for the short form. Participants were asked to consider their experiences over the past two weeks when completing the scale. The 7 items in the WEMWBS-SF are more closely related to functioning than to emotions. The validity and reliability of the WEMWBS-SF were examined in a sampl
Quality of Life Score | Assessments will be conducted at three time points: baseline, post-intervention (after 7 weeks), and at the 19-week follow-up.
  The World Health Organization Quality of Life-BREF (WHOQOL-BREF) is a 26-item abbreviated version of the 100-item World Health Organization Quality of Life Assessment (WHOQOL), designed to evaluate an individual's perception of their quality of life. The scale is composed of four domains: general health, physical health, social relationships, and environment. The Turkish adaptation of the WHOQOL-BREF was conducted by Eser et al. (1999). The scale does not have a fixed total score; rather, an increase in score indicates an improvement in perceived quality of life.
General Self-Efficacy Score | Assessments will be conducted at three time points: baseline, post-intervention (after 7 weeks), and at the 19-week follow-up.
  Originally developed in Germany in 1979 by Jerusalem and Schwarzer, the scale initially consisted of 20 items. In 1981, the same researchers revised the scale, reducing it to 10 items. In subsequent years, this four-point Likert-type scale (completely false = 1, completely true = 4) has been translated into numerous languages, and its validity and reliability have been extensively studied. Kaiser-Guttman eigenvalue and scree plot analyses have consistently indicated a single-factor solution across different countries. Subsequently, confirmatory factor analysis was conducted to test both one-factor and two-factor models. The results of confirmatory factor analysis supported the assumption of a single-factor structure. All items on the scale are positively scored, with a possible range of 10 to 40 points, and higher scores indicate higher levels of general self-efficacy. The Turkish adaptation and validation of the scale were conducted by Apay (2010).
Self-Esteem Score | Assessments will be conducted at three time points: baseline, post-intervention (after 7 weeks), and at the 19-week follow-up.
  Developed by Rosenberg in 1965, the Rosenberg Self-Esteem Scale is a self-report measure originally composed of 63 multiple-choice items, divided into 12 subscales. For the purpose of measuring self-esteem, the first 10 items were selected for this study. Çuhadaroğlu (1986) conducted a Turkish adaptation and validation study, reporting a Cronbach's alpha of 0.81. The scale employs a four-point Likert format (strongly agree, agree, disagree, strongly disagree). Scoring involves assigning 4 points for "strongly agree" on positive items and 1 point for "strongly disagree," with the reverse scoring for negative items. The total score is calculated by summing the scores of the 10 items and dividing by 10. A higher average score indicates higher self-esteem.
Visual Analog Scale for Anxiety | Assessments will be conducted at three time points: baseline, post-intervention (after 7 weeks), and at the 19-week follow-up.
  The Visual Analog Scale for Anxiety (VAS-A) is a simple yet effective method for assessing anxiety levels in patients. By providing a continuous 10 cm scale anchored by "no anxiety" and "highest possible anxiety," the VAS-A allows patients to subjectively rate their current anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Kilis 7 Aralık Üniversitesi, Kilis, Kilis, Turkey (Türkiye)